CLINICAL TRIAL: NCT00307398
Title: Anecortave Acetate Risk-Reduction Trial (AART)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Management decision
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-02-60
Record Dates: First submitted 2006-03-24; First posted 2006-03-28 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2009-05

CONDITIONS: Dry AMD
Keywords: AMD; Dry AMD; Drusen; CNV
MeSH Terms: interventions — anecortave acetate; AL 3789

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- AL-3789 (Experimental): One injection to the study eye by the posterior juxtascleral depot procedure at 6-month intervals for 42 months.
  Interventions: Drug: Anecortave Acetate (AL-3789) sterile suspension, 15 mg or 30 mg
- Anecortave Acetate Vehicle (Sham Comparator): One sham injection to the study eye at 6-month intervals for 42 months. Syringe containing AA vehicle was not inserted into the eye.
  Interventions: Other: Anecortave Acetate Vehicle

INTERVENTIONS:
Drug: Anecortave Acetate (AL-3789) sterile suspension, 15 mg or 30 mg — One 0.5 mL injection of 30 mg/mL (AA 15 mg) or one 0.5 mL injection of 60 mg/mL (AA 30 mg) into a posterior juxtascleral depot (PJD) at 6-month intervals.
  Arms: AL-3789
Other: Anecortave Acetate Vehicle — One 0.5 mL sham injection at 6-month intervals. Syringe containing AA vehicle was not inserted into the eye.
  Arms: Anecortave Acetate Vehicle

SUMMARY:
A 48 month study of posterior juxtascleral administrations of Anecortave Acetate 15 or 30 mg or sham administration every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Dry AMD study eye, Wet AMD non-study eye.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Age
* Other protocol-defined exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2596 (Actual)
Dates: Start 2004-03; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with sight-threatening choroidal neovascularization (ST-CNV) in the study eye at Month 48 | Month 48
  ST-CNV is defined as CNV or a portion of CNV within 2500 microns of the foveal center, as evidenced by digital angiography at the clinical site.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Zilliox, Study Director — Study Manager
Locations (1):
- Study Centers in the United States and Globally, Fort Worth, Texas, United States